CLINICAL TRIAL: NCT06381258
Title: Fetal Systolic and Diastolic Cardiac Function Assessment in Mothers with Preeclampsia
Brief Title: Fetal Cardiac Function
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer of Obs& Gyn. Specialist of Urogynecology, Assiut University
Other Study IDs: SDF
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-04

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with preeclampsia: Fetal ultrasound( echocardiography).Measurements will be performed using conventional pulsed-wave Doppler and M mode cross sectional image of the fetal thorax at the level of the 4-chamber view with an apical projection of the heart is obtained. Measurements of the ventricle at diastole and systole are obtained, and using the relationship between these measurements, calculations are performed to determine the ejection fraction (EF) ([diastole measurement-systole measurement]/diastole) measurement and shortening fraction ( SF) for both right & left ventricles.
  Assessment of ventricular diastolic function through measuring E-wave (early ventricular filling) and A wave (active atrial contraction - late ventricular filling) peak velocities and the ratio between them (E/A ratio) as an index will be performed for both mitral valve (MV) and tricuspid valve (TV)
  Interventions: Procedure: Ultrasound
- Patients without preeclampsia: Fetal ultrasound (echocardiography).Measurements will be performed using conventional pulsed-wave Doppler and M mode cross sectional image of the fetal thorax at the level of the 4-chamber view with an apical projection of the heart is obtained. Measurements of the ventricle at diastole and systole are obtained, and using the relationship between these measurements, calculations are performed to determine the ejection fraction (EF) ([diastole measurement-systole measurement]/diastole) measurement and shortening fraction ( SF) for both right & left ventricles.
  Assessment of ventricular diastolic function through measuring E-wave (early ventricular filling) and A wave (active atrial contraction - late ventricular filling) peak velocities and the ratio between them (E/A ratio) as an index will be performed for both MV and TV
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Fetal echocardiography using ultrasound device

SUMMARY:
The aim of our study is to evaluate the effect of PE and FGR on fetal cardiac function. Pregnancies with preeclampsia and FGR, and preeclampsia with normal fetal growth are evaluated by echocardiography and compared with uncomplicated pregnancies.

DETAILED DESCRIPTION:
Preeclampsia (PE) represent a major concern in public health, affecting 2-8% of all pregnancies and considered one of the leading causes of perinatal morbidity and mortality. Fetal growth restriction (FGR) ia also a common health problem affecting about 5-10% of all pregnancies and commonly associates with preeclampsia . It is estimated that 20% of cases of PE present with FGR and about 50% of early-onset FGR cases will eventually coexist with PE .

Both syndromes share some pathophysiologic features, with a variable involvement of placental insufficiency and cause fetal cardiovascular remodeling and adaptations . Fetal adaptations as metabolic and cardiovascular programming occur in response to adverse intrauterine conditions as PE and FGR . Offspring from preeclamptic pregnancies showed cardiac structural and functional changes and greater blood pressure in childhood and adolescence .

Most of the studies on FGR included pregnancies complicated by PE and vice versa, which fails to adequately assess the independent effect of each condition on the fetal cardiac functions.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women more than or equals 28 weeks
* Preeclampsia defined as systolic blood pressure 140 mm Hg and/or diastolic blood pressure 90 mm Hg
* Fetus with normal growth or with growth restriction

Exclusion criteria:

* congenital malformations
* intrauterine infection
* multiple pregnancies
* fetuses of mothers treated with a tocolytic agent
* fetuses with abnormal heart rates (tachycardia or bradycardia)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group A : patients with preeclampsia (either with FGR or normal growth) Group B : patients without preeclampsia (16 cases)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Cardiac systolic function | 4 months
  Measurement of ejection fraction in percent % (high is good, low is bad)

SECONDARY OUTCOMES:
Cardiac diastolic function | 4 months
  Measurement of spherity index ( high is bad, low is good)

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No